CLINICAL TRIAL: NCT06296160
Title: Role of Lung Ultrasound in the Assessment and Management of Pulmonary Congestion in Chronic Hemodialysis Patients: A Randomized Controlled Study
Brief Title: A Simplified Lung Ultrasound Guided Management Protocol Of Pulmonary Congestion in Hemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Abdullah Ibrahim Hamad, Lead Principal Investigation, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MRC-01-23-035; LUSAM-HD (Other Grant/Funding Number: COMITE D'ETHIQUE du CHU BRUGMANN c/o Direction Médicale)
Record Dates: First submitted 2024-02-18; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: End Stage Renal Disease
Keywords: Regular Hemodialysis; Fluid overload; lung cognition; Number of B-lines; Lung Ultrasound
MeSH Terms: conditions — Kidney Failure, Chronic; Edema

STUDY DESIGN:
Intervention Model Description: The study will compare two groups according to the dry weight determination method:
  (1) Control arm- modification of dry weight according to standardized care only. The standard of care to modify dry weight is what nephrologists use actually to define the best theoretical dry weight, including clinical (blood pressure, edema, shortness of breath, lung auscultation, etc.) and laboratory measures (Protein concentration before and after dialysis sessions …). (2) Intervention arm- modify patient's dry weight according to standard of care + B lines score on lung ultrasound BLS obtained after the midweek dialysis session, considered as Day one (Day 1)
Who Masked: Participant
Masking Description: It is a single-blinded trial as the treatment is blinded by Subjects only, meaning that the type of dry weight modification will not be disclosed to the subject, and they will not know which group he/she will be in at the time of consenting to limit the bias in opinion. The investigator and the research team must know the type of treatment, as the investigator will modify the dry weight according to the treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Based on the Ultrasound result, Dry Weight Modification:
  Duration: 2 months. Number of visits: 5 visits.
  A- Intervention Phase (Dry weight modification)= [Day-1 and Day-15]
  B- Observational Phase (No Dry weight modification on Day 30, Day 45, and Day 60).
  Interventions: Other: Intervention Group
- Control Arm (No Intervention): * Includes patients who will receive usual ambulatory and at-discharge care.
  * No dry-weight modification (The study investigators will not modify the dry weight).
  * All subjects in the Control group will be under follow-up close observation for two months [5 visits].
  * The participant will follow the standard of care practice (Dry Weight evaluation according to clinical judgment by the assigned physician and biological data.
  Study procedures:
  1. Obtain a lung ultrasound after the midweek dialysis session.
  2. The 8-zone lung ultrasound method calculates the number of B-line scores.
  3. Check the Blood Pressure 3 times/day on non-Dialysis days.
  4. Check the ambulatory blood pressure for 48 hours (Baseline on Day 1 and Follow-up on Day 60).

INTERVENTIONS:
Other: Intervention Group — A- (Intervention Phase= (Day-1) + (Day-15)
  1. Obtain a lung ultrasound after the midweek dialysis session.
  2. The 8-zone lung ultrasound method calculates the number of B-line scores.
  3. Reduce the dry weight by 500 g if the B-line score is >0.54/zone (BLS>5). considered a day one.
  4. The dry weight will be reduced only if the arterial blood pressure at the end of the session is BP >110/60 mmHg and the patient had no hypotension episode during the session.
  5. The adjustment of dry weight based on lung ultrasound should not be made on the same day as the standard approach adjustment (Regular monthly clinical standards modification.
  6. Check the Blood Pressure 3 times/ day on the non-dialysis following the ultrasound.
  7. Check the ambulatory blood pressure for 48 hours (Baseline on day 1 and Follow-up on Day 60).
  B - Observational Phase= (Day-30) + (Day-45) + (Day-60)].
  Other Names: Dry- Weight modification
  Arms: Interventional Arm

SUMMARY:
Pulmonary congestion secondary to volume overload or interstitial tissue inflammation is common in chronic hemodialysis patients. This pulmonary congestion occurs mainly during the period between dialysis sessions and is an independent risk factor for cardiovascular event morbidity and mortality in this population. The evaluation of this pulmonary congestion and the estimation of the dry weight of hemodialysis patients according to conventional methods represent a real challenge for clinical nephrologists. Lung ultrasound is a new diagnostic approach validated in the assessment of pulmonary congestion. It would allow a better assessment of dry weight in chronic hemodialysis patients based on the results of preliminary studies, including our latest pilot study. However, there is little evidence comparing this novel approach to traditional approaches.

DETAILED DESCRIPTION:
The classic treatment program for hemodialysis patients includes three sessions per week on fixed days (Monday-Wednesday-Friday or Tuesday-Thursday-Saturday or Sunday).

Hemodialysis patients with end-stage renal disease often develop fluid overload between dialysis sessions due to decreased diuresis or anuria. This overload is manifested by pulmonary congestion, which is an independent risk factor for morbidity and mortality from cardiovascular events in these patients. Studies show pulmonary congestion is not always associated with increased left ventricular filling pressure. Patients with end-stage renal disease also have impaired capillary permeability secondary to the dialysis filters used (synthetic membranes) and uremic syndromes, which increases their risk of cardiopulmonary complications. In addition, some experimental studies show that inflammatory mechanisms can also cause capillary changes and increase the risk of pulmonary edema in patients with end-stage renal disease with fluid overload. Evaluating fluid overload and estimating the dry weight of hemodialysis patients.

According to conventional methods, namely pulmonary auscultation, chest radiography, cardiac ultrasound, and blood pressure measurement, this represents a real challenge for clinical nephrologists. Hyper- or hypo-hydration in hemodialysis patients, especially if it persists over time, is linked to adverse cardiovascular consequences. The investigators currently know that this increase in extravascular fluid in the lungs creates an air-liquid interface that induces an ultrasound artifact in continuous lines called B-lines, which ultrasound machines can detect. It has been shown that the presence of these B-lines alone in hemodialysis patients is an independent risk factor for mortality and cardiovascular events. Their sensitivity is high and can be detected even at the subclinical stage. Similarly, in hemodialysis patients with high blood pressure, the modification of dry weight according to these B-lines has demonstrated a beneficial effect on blood pressure control and cardiac parameters. It should be noted that these B-lines are not specific for water overload and can be the consequence of several pathologies, such as interstitial pneumonia or diffuse pulmonary fibrosis. Lung ultrasound is a new diagnostic approach validated in the assessment of pulmonary congestion. According to recent preliminary reports, it would allow a better estimate of volume expansion and, therefore, a better assessment of dry weight in chronic hemodialysis patients. However, little evidence compares this novel approach to conventional standardized approaches. No study has defined the best moment to do a lung ultrasound to obtain the most reliable pulmonary congestion level. The investigators did this in our pilot study and concluded that the best moment was after the second dialysis session. Based on that, and in order to establish a management and monitoring protocol, the study aimed to show that reducing dry weight. According to lung ultrasound at that particular moment, it is the best way to manage pulmonary congestion in this population. Dialysis service in Qatar is provided by Hamad Medical Corporation facilities. The investigators have seven units providing ambulatory dialysis care. Currently, The investigators have about 1000 hemodialysis (HD) patients.

The largest center with over 500 patients is Fahad Bin Jassim Kidney Center (FBJKC). Our current practice is to estimate dry weight on a monthly basis during the monthly evaluation of HD patients by our nephrologist. This evaluation depends on physical examination, blood pressure, and other clinical parameters. Sometimes, it is very difficult to estimate the dry weight (obesity, bedbound or wheelchair-dependent patients, congestive heart failure, etc.). Introducing new technology to guide the estimation of dry weight provides great service to our HD patients. It can help in estimating dry weight, especially in difficult cases. Lung ultrasound to evaluate congestion is a newly introduced technology to help estimate dry weight. Implementing this technology might offer valued service to improve care to our HD patients in Qatar. I want to highlight the importance of this study to our dialysis service in Qatar. In addition to the specified novel approach mentioned in the methods and outcomes, the investigators have many goals to serve dialysis services in Qatar. The investigators will introduce Lung US volume assessment (currently not done) with the training needed and validate the best way of utilizing it to serve our patients. The investigators will also introduce ambulatory home blood pressure measurement (currently not done in dialysis) with all the training needed for our service and the best way to apply it. This study has scientific and practical values on the research ground with the expected immediate impact on our dialysis service.

ELIGIBILITY:
Inclusion Criteria:

* Chronic in-center hemodialysis patients for at least three months

Exclusion Criteria:

* Active Cancer.
* Active infection.
* Patients with pulmonary fibrosis.
* Patients with diffuse pneumonia.
* Patients with frequent hypotension episodes in HD
* Extreme weight gain between dialysis sessions demanding more than 13 ml/kg/h UF rate.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of adding B-line score evaluation through lung ultrasound to the standard of care to improve pulmonary congestion (measured by B lines score) in hemodialysis patients | At baseline and at the end of 2 months follow-up
  Comparing the difference in B lines score (that reflects lung congestion) between both groups before (LUS day 1) and after (LUS day 60) the intervention (fluid removal adjustment by changing dry weight). B-line score is >0.54/zone (BLS>5) is cut-off score. 0-5 B-lines (BLS≤5) indicate [No- Mild lung Congestion], and if B-lines more than (BLS>5) lines; indicate [Moderate-severe lung congestion].

SECONDARY OUTCOMES:
The impact of utilizing B lines score based additional fluid removal on interdialytic ambulatory blood pressure. | At baseline and at the end of 2 months follow-up
  Interdialytic blood pressure
The impact of utilizing B lines score based additional fluid removal on intradialytic ambulatory blood pressure | At baseline and at the end of 2 months follow-up
  1. 24-hour ambulatory blood pressure measurement (ABPM) for 44H at day -2 and day 28.
  2. Ambulatory home blood pressure by using a standard blood pressure machine at days (2, 9, 16, 23, 31)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Al-Malki, MD, Study Director — Hamad Medical Corporation
Locations (1):
- Kaysi Saleh, Brussels, Van Gehuchten, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The coded master sheet with all the subject medical history and the lung US results will be sent to the Belgium site through DropBox, which is a secure server for data storage and transferring to ensure the security of the data, it has a partnership with Microsoft, which allows synchronization speed for large files that improve the upload or download time between the two sites.
Supporting Information: CSR
Time Frame: Every six months.
Access Criteria: through DropBox, which is a secure server for data storage and transferring to ensure the security of the data, it has a partnership with Microsoft, which allows synchronization speed for large files that improve the upload or download time between the two sites.

REFERENCES:
- [Result] Shoji T, Tsubakihara Y, Fujii M, Imai E. Hemodialysis-associated hypotension as an independent risk factor for two-year mortality in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1212-20. doi: 10.1111/j.1523-1755.2004.00812.x. PMID 15327420
- [Result] Zoccali C, Torino C, Tripepi R, Tripepi G, D'Arrigo G, Postorino M, Gargani L, Sicari R, Picano E, Mallamaci F; Lung US in CKD Working Group. Pulmonary congestion predicts cardiac events and mortality in ESRD. J Am Soc Nephrol. 2013 Mar;24(4):639-46. doi: 10.1681/ASN.2012100990. Epub 2013 Feb 28. PMID 23449536
- [Result] Torino C, Gargani L, Sicari R, Letachowicz K, Ekart R, Fliser D, Covic A, Siamopoulos K, Stavroulopoulos A, Massy ZA, Fiaccadori E, Caiazza A, Bachelet T, Slotki I, Martinez-Castelao A, Coudert-Krier MJ, Rossignol P, Gueler F, Hannedouche T, Panichi V, Wiecek A, Pontoriero G, Sarafidis P, Klinger M, Hojs R, Seiler-Mussler S, Lizzi F, Siriopol D, Balafa O, Shavit L, Tripepi R, Mallamaci F, Tripepi G, Picano E, London GM, Zoccali C. The Agreement between Auscultation and Lung Ultrasound in Hemodialysis Patients: The LUST Study. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):2005-2011. doi: 10.2215/CJN.03890416. Epub 2016 Sep 22. PMID 27660305
- [Result] Maw AM, Hassanin A, Ho PM, McInnes MDF, Moss A, Juarez-Colunga E, Soni NJ, Miglioranza MH, Platz E, DeSanto K, Sertich AP, Salame G, Daugherty SL. Diagnostic Accuracy of Point-of-Care Lung Ultrasonography and Chest Radiography in Adults With Symptoms Suggestive of Acute Decompensated Heart Failure: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Mar 1;2(3):e190703. doi: 10.1001/jamanetworkopen.2019.0703. PMID 30874784
- [Result] Zoccali C, Tripepi R, Torino C, Bellantoni M, Tripepi G, Mallamaci F. Lung congestion as a risk factor in end-stage renal disease. Blood Purif. 2013;36(3-4):184-91. doi: 10.1159/000356085. Epub 2013 Dec 20. PMID 24496189
- [Result] Reisinger N, Lohani S, Hagemeier J, Panebianco N, Baston C. Lung Ultrasound to Diagnose Pulmonary Congestion Among Patients on Hemodialysis: Comparison of Full Versus Abbreviated Scanning Protocols. Am J Kidney Dis. 2022 Feb;79(2):193-201.e1. doi: 10.1053/j.ajkd.2021.04.007. Epub 2021 Jun 3. PMID 34090905
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Saad MM, Kamal J, Moussaly E, Karam B, Mansour W, Gobran E, Abbasi SH, Mahgoub A, Singh P, Hardy R, Das D, Brown C, Kapoor M, Demissie S, Kleiner MJ, El Charabaty E, El Sayegh SE. Relevance of B-Lines on Lung Ultrasound in Volume Overload and Pulmonary Congestion: Clinical Correlations and Outcomes in Patients on Hemodialysis. Cardiorenal Med. 2018;8(2):83-91. doi: 10.1159/000476000. Epub 2017 Nov 29. PMID 29617006
- [Result] Loutradis C, Papadopoulos CE, Sachpekidis V, Ekart R, Krunic B, Karpetas A, Bikos A, Tsouchnikas I, Mitsopoulos E, Papagianni A, Zoccali C, Sarafidis P. Lung Ultrasound-Guided Dry Weight Assessment and Echocardiographic Measures in Hypertensive Hemodialysis Patients: A Randomized Controlled Study. Am J Kidney Dis. 2020 Jan;75(1):11-20. doi: 10.1053/j.ajkd.2019.07.025. Epub 2019 Nov 12. PMID 31732234
- [Result] Loutradis C, Sarafidis PA, Ekart R, Papadopoulos C, Sachpekidis V, Alexandrou ME, Papadopoulou D, Efstratiadis G, Papagianni A, London G, Zoccali C. The effect of dry-weight reduction guided by lung ultrasound on ambulatory blood pressure in hemodialysis patients: a randomized controlled trial. Kidney Int. 2019 Jun;95(6):1505-1513. doi: 10.1016/j.kint.2019.02.018. Epub 2019 Mar 5. PMID 31027889
- [Result] Hoke TS, Douglas IS, Klein CL, He Z, Fang W, Thurman JM, Tao Y, Dursun B, Voelkel NF, Edelstein CL, Faubel S. Acute renal failure after bilateral nephrectomy is associated with cytokine-mediated pulmonary injury. J Am Soc Nephrol. 2007 Jan;18(1):155-64. doi: 10.1681/ASN.2006050494. Epub 2006 Dec 13. PMID 17167117
- [Result] K/DOQI Workgroup. K/DOQI clinical practice guidelines for cardiovascular disease in dialysis patients. Am J Kidney Dis. 2005 Apr;45(4 Suppl 3):S1-153. No abstract available. PMID 15806502
- [Result] Assimon MM, Wenger JB, Wang L, Flythe JE. Ultrafiltration Rate and Mortality in Maintenance Hemodialysis Patients. Am J Kidney Dis. 2016 Dec;68(6):911-922. doi: 10.1053/j.ajkd.2016.06.020. Epub 2016 Aug 26. PMID 27575009
- [Result] Kim TW, Chang TI, Kim TH, Chou JA, Soohoo M, Ravel VA, Kovesdy CP, Kalantar-Zadeh K, Streja E. Association of Ultrafiltration Rate with Mortality in Incident Hemodialysis Patients. Nephron. 2018;139(1):13-22. doi: 10.1159/000486323. Epub 2018 Jan 18. PMID 29402814
- [Result] Flythe JE, Kimmel SE, Brunelli SM. Rapid fluid removal during dialysis is associated with cardiovascular morbidity and mortality. Kidney Int. 2011 Jan;79(2):250-7. doi: 10.1038/ki.2010.383. Epub 2010 Oct 6. PMID 20927040
- [Result] Loutradis C, Sarafidis PA, Ekart R, Tsouchnikas I, Papadopoulos C, Kamperidis V, Alexandrou ME, Ferro CJ, Papagianni A, London G, Mallamaci F, Zoccali C. Ambulatory blood pressure changes with lung ultrasound-guided dry-weight reduction in hypertensive hemodialysis patients: 12-month results of a randomized controlled trial. J Hypertens. 2021 Jul 1;39(7):1444-1452. doi: 10.1097/HJH.0000000000002818. PMID 34074973
- [Derived] Kaysi S, Hamad A, Boulgheraif A, Bonkain F, Libertalis M, Abu Ayyach A, Baz M, Farah I, Ibrahim R, Ateya H, Mathew M, Collart F, Mesquita M, Taghavi M, Alkadi M, Al-Malki H, Nortier J. Lung Ultrasound Guided Management of Pulmonary Congestion in Hemodialysis: A Multicenter Randomized Controlled Trial. Kidney360. 2026 Jan 1;7(1):139-149. doi: 10.34067/KID.0000000873. Epub 2025 Aug 15. No abstract available. PMID 40815555